CLINICAL TRIAL: NCT06510218
Title: The 2021-2022 Study of Family and Staff Well-Being in Head Start AIAN FACES Programs
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 51307-B
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Head Start Participation
Keywords: child care; child development; child health; child rearing; children; curriculum; early childhood education; families; Head Start; parenting; parents; parent well-being; teacher well-being; early childhood workforce; school readiness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head Start children and families: Children (261) Parents (261) Teachers (88) Program directors (18) Center directors (43)

SUMMARY:
The 2021-2022 Study of Family and Staff Experiences in American Indian and Alaska Native Head Start Family and Child Experiences Survey Programs (the 2021-2022 Study) builds on AIAN FACES 2019, a national study of children and families participating in Head Start programs funded through grants to federally recognized tribes and consortia. In the year following the start of the COVID-19 pandemic, there was a need to understand how children, families, and Head Start staff were faring. The 2021-2022 Study explores this with some of the programs that participated in AIAN FACES 2019.

DETAILED DESCRIPTION:
The American Indian and Alaska Native Head Start Family and Child Experiences Survey (AIAN FACES) provides information about children and families enrolled in Head Start programs operated by federally recognized tribes (known as Region XI AIAN Head Start). Nationally representative studies were conducted in the 2015-2016 and 2019-2020 program years (entered as NCT03842111 and NCT04046965, respectively).

The motivation and goals of the 2021-2022 Study of Family and Staff Experiences in AIAN FACES Programs came from a need to learn about children's, families', and teachers' experiences as the COVID-19 pandemic continued affecting Region XI Head Start families' and staff's lives into another program year-and from recognizing the disproportionate impact of the pandemic on AIAN communities. The Office of Planning, Research, and Evaluation in the Administration for Children and Families (ACF), U.S. Department of Health and Human Services, funded Mathematica to conduct a new data collection effort, the 2021-2022 Study, for the fall and spring of the 2021-2022 program year. The goals were to provide data on the characteristics and needs of Region XI children, families, and staff starting 18 months into the COVID-19 pandemic, and to provide information to help better understand staff retention and turnover.

The 2021-2022 Study includes data from a multistage sample of Region XI Head Start programs (based on the AIAN FACES 2019 sample), centers, teachers, and families from across the United States. Data from the 2021-2022 Study provide a window into the experiences of a small number of Region XI children, their families, and staff who were able to participate in data collection between October 2021 and July 2022. The data do not represent all Region XI Head Start children, their families, and staff nationally. They provide a snapshot of the experiences of children in Region XI Head Start children, their families, and staff during this difficult time.

ELIGIBILITY:
Inclusion Criteria: The Head Start programs participating in the 2021-2022 Study were a probability sample selected from among 146 study-eligible programs on the 2016-2017 Head Start Program Information Report (PIR). To be eligible for the study, a program had to be

* providing services directly to children ages 3 to 5

  o The Head Start Program Performance Standards require that children turn 3 by date used to determine eligibility for public school in the community in which the Head Start program is located. Therefore, some study children were 2 years old at the time of sampling if sampling occurred before the date used for public school eligibility.
* not be in imminent danger of losing its grantee status. Probability samples of centers were selected within each program, teachers within each center, and children within each teacher. Further, the programs that participated in the 2019-2020 study had to have participated in AIAN FACES 2019-2020.

Exclusion Criteria: Head Start programs in Regions I through X and Migrant and Seasonal Head Start (Region XII) were not eligible for the 2021-2022 Study. Programs that did not participate in AIAN FACES 2019-2020 were also not eligible for this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Region XI Head Start children (and their families), Region XI Head Start programs, Region XI Head Start centers, Region XI Head Start classrooms/teachers.
Sampling Method: Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
General health status | October 2021-January 2022; April-July 2022
  Indicators of physical well-being were assessed by parent report to a survey item on if child's health is excellent, very good, good, fair, or poor
Social-emotional development | November 2021-January 2022; April-July 2022
  Indicators of social-emotional development were assessed using teacher report of several items on children's positive and problem behaviors. Please see the 2021-2022 Study User's Manual (Reid et al. 2024) for more information on the scores and technical information.
Social-emotional development - Approaches to learning | October 2021-January 2022; April-July 2022
  Indicators of social-emotional development were assessed using teacher and parent report of approaches to learning using the Early Childhood Longitudinal Study - Kindergarten Class of 1998 (ECLS-K). The items assess a child's motivation, attention, organization, persistence, and independence in learning. Please see U.S. Department of Education 2002 for more information on the scores and technical properties.
Parents' depressive symptoms | October 2021-January 2022; April-July 2022
  Parents' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Teachers' depressive symptoms | November 2021-January 2022; April-July 2022
  Teachers' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Program directors' depressive symptoms | April-July 2022
  Program directors' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Center directors' depressive symptoms | April-July 2022
  Center directors' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Parents' anxiety | October 2021-January 2022; April-July 2022
  Parents' and caregivers' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Teachers' anxiety | November 2021-January 2022; April-July 2022
  Teachers' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Program directors' anxiety | April-July 2022
  Program directors' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Center directors' anxiety | April-July 2022
  Center directors' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Staffing challenges | April-July 2022
  Staffing challenges were measured by summarizing center director survey items about the extent to which staff turnover has been a problem in terms of maintaining consistency in operations and care of children, and about finding classroom coverage and having enough staff to operate at full capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bernstein, Ph.D., Study Director — Mathematica Policy Research, Inc.; Nikki Aikens, Ph.D., Principal Investigator — Mathematica Policy Research, Inc.; Louisa Tarullo, Ed.D., Principal Investigator — Mathematica Policy Research, Inc.; Ashley Kopack Klein, M.A., Study Director — Mathematica Policy Research, Inc.
Locations (1):
- Mathematica, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
In the future, the 2021-2022 Study of Family and Staff Experiences in AIAN Head Start FACES Programs archived data will be available for access.
Time Frame: Data will become available within 2 years of completion.
Access Criteria: Applications for access to restricted-use data file will include completing and adhering to a User Agreement, and undergoing review by the AIAN FACES Data Committee.

REFERENCES:
- [Background] Radloff, L. "The CES-D Scale: A Self-Report Depression Scale for Research in the General Population." Applied Psychological Measurement, vol. 1, no. 3, 1977, pp. 385-401.
- [Background] Reid, M., A. Kopack Klein, E. Doran, B. Lepidus Carlson, J. Cannon, N. Aikens, N. Reid, S. Skidmore, K. Gonzalez, X. Li, L. Malone, S. Bernstein. "2021-2022 Study of Family and Staff Experiences in AIAN Head Start FACES Programs (2021-2022 Study): User's Manual." Washington, DC: Mathematica, 2024.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] U.S. Department of Education, National Center for Education Statistics. Early Childhood Longitudinal Study-Kindergarten Class of 1998-99 (ECLS-K), Psychometric Report for Kindergarten through First Grade. NCES 2002-05. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2002.